CLINICAL TRIAL: NCT02524561
Title: KEEPS Mammographic Density And Breast Health Ancillary Study
Acronym: KEEPS MDBHAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Kronos Longevity Research Institute (Other); Albert Einstein College of Medicine (Other); Columbia University (Other); Mayo Clinic (Other); University of California, San Francisco (Other); University of Utah (Other); University of Washington (Other); Yale University (Other)
Responsible Party: Principal Investigator, Rulla Tamimi, Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2009P002326; R01CA136918 (NIH)
Record Dates: First submitted 2015-08-13; First posted 2015-08-17 (Estimated); Results first posted 2017-03-08 (Actual); Last update posted 2017-03-08 (Actual); Status verified 2017-01

CONDITIONS: Mammographic Density; Abnormal Mammogram
Keywords: mammographic density; abnormal mammogram; biopsy
MeSH Terms: interventions — 2-chloroethyl ethyl sulfide; Estrogens, Conjugated (USP); Ortho Evra; Estradiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CEE pill, active progesterone (Active Comparator): Conjugated equine estrogens 0.45 mg/day, placebo patch, Prometrium (micronized progesterone USP encapsulated with peanut oil) 200 mg daily for the first 12 days of each month at bedtime
  Interventions: Drug: CEE pill; Drug: Active Progesterone; Other: Placebo patch
- estradiol patch, active progesterone (Active Comparator): Transdermal estradiol, 50 mcg/day, placebo tablet, Prometrium (micronized progesterone USP encapsulated with peanut oil) 200 mg daily for the first 12 days of each month at bedtime
  Interventions: Drug: Estradiol patch; Drug: Active Progesterone; Other: Placebo tablet
- placebo (Placebo Comparator): Placebo tablet, placebo patch, placebo progesterone
  Interventions: Other: Placebo tablet; Other: Placebo patch; Other: Placebo progesterone

INTERVENTIONS:
Drug: CEE pill — Conjugated equine estrogens 0.45 mg/day
  Other Names: premarin
  Arms: CEE pill, active progesterone
Drug: Estradiol patch — Climara 50 mcg/day
  Other Names: Climara 50 mcg/day
  Arms: estradiol patch, active progesterone
Drug: Active Progesterone — Prometrium (micronized progesterone USP encapsulated with peanut oil) 200 mg daily for the first 12 days of each month at bedtime
  Arms: CEE pill, active progesterone; estradiol patch, active progesterone
Other: Placebo tablet — Placebo tablet
  Arms: estradiol patch, active progesterone; placebo
Other: Placebo patch — placebo patch
  Arms: CEE pill, active progesterone; placebo
Other: Placebo progesterone — placebo progesterone
  Arms: placebo

SUMMARY:
Combined estrogen and progestin therapy has been shown to increase mammographic density and incidence of breast cancer in randomized trials. The investigators propose to examine the effects of now commonly used low-dose combined hormone therapy (HT) regimens on breast density, rates of abnormal mammogram, and circulating estrogens in the ongoing, already-funded Kronos Early Estrogen Prevention Study (KEEPS). KEEPS is a randomized clinical trial with a primary goal of examining the effects of low-dose transdermal versus oral estrogen combined with cyclic micronized progesterone on progression of subclinical atherosclerosis in recently menopausal women. Prior studies of low-dose HT have been of short duration and small size. By determining the effects of low-dose hormone therapy on the breast, the proposed ancillary study will add important information about the estimated balance of risks and benefits associated with low-dose HT and will help guide future research trials.

DETAILED DESCRIPTION:
Despite data from clinical trials showing an increased risk of breast cancer and lack of overall benefit for primary prevention with hormone therapy (HT), there is still significant usage of HT by clinicians and women for treatment of moderate-to-severe systemic menopausal symptoms. Due to the possible increased risks with these preparations, current clinical recommendations advocate utilizing the lowest dose for the shortest possible duration, but average duration is often for 2-4 years. However, the effects of commonly used low-dose HT regimens on breast density and breast cancer risk are unknown. Recent data from intervention trials support the long standing hypothesis that hormonal effects on breast cancer risk are mediated through breast density. The Kronos Early Estrogen Prevention Study (KEEPS) is an ongoing, already- funded randomized clinical trial with a primary goal of examining the effects of 4 years of low- dose transdermal versus oral estrogen combined with cyclic micronized progesterone on progression of subclinical atherosclerosis in recently menopausal women. The proposed ancillary study will efficiently examine the effects of randomized low-dose HT on key breast cancer surrogate endpoints: mammographic density and rates of abnormal mammograms. In the parent KEEPS study, a total of 720 women were randomized to oral conjugated equine estrogens (0.45 mg/d), transdermal 17-beta estradiol (50 mcg/d), or placebo, with cyclic micronized progesterone (200 mg for 12 days) for active hormonal therapy groups. All participants were required to have mammography prior to study entry as well as yearly during follow-up; blood samples also were collected at these time points. Randomization was completed in 2008. In this ancillary study, we aimed to collect mammograms from eligible women consenting to be part of the ancillary study(n=517) from baseline, year 1 and year 3 will be obtained and processed centrally to calculate mammographic density. The investigators will determine if these two low-dose HT regimens are associated with change in mammographic density. The investigators will also examine if baseline mammographic density or circulating biomarkers including estradiol, estrone, and estrone sulfate, modify or mediate changes in breast density with HT. In addition, the effects of hormonal regimens on the rates of abnormal mammogram and biopsy will be determined. By determining the effects of low-dose combined HT on the breast, the proposed study will add timely and important information about the estimated balance of risks and benefits associated with low-dose HT and will help guide future research.

ELIGIBILITY:
Inclusion Criteria:

* Women were 42-58 years of age, have had cessation of menses at or after age 40 and no menses for a minimum of 6 and a maximum of 36 months at screening.
* Subjects may or may not have had current vasomotor estrogen deficiency symptoms, had not taken estrogen- or progestogen-containing medication (oral contraceptive or hormone replacement) within 3 months of randomization, and had plasma FSH levels measured at ≥35 ng/ml and plasma E2 levels of <40 pg/ml.

Exclusion Criteria:

* Subjects were excluded for increased endometrial thickness on ultrasound >5 mm, unless endometrial biopsy was negative; for LDL ≥ 190 mg/dl or triglycerides ≥ 400 at screening, or use of lipid lowering drugs.

Ages: 42 Years to 58 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 517 (Actual)
Dates: Start 2005-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Rexrode, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
We are willing to share data with collaborators if analyses are approved by the investigative team and approved by our IRB.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women in the parent study were approached to be part of this ancillary study (MDBHAS). For women who consented we attempted to collect their mammograms. Our collection took place after they started and were randomized in the parent study.
Period: Baseline: Pre-randomization Mammogram
Arm/Group | CEE Pill, Active Progesterone | Estradiol Patch, Active Progesterone | Placebo
Started | 168 (Consented to MDBHAS) | 162 (Consented to MDBHAS) | 187 (Consented to MDBHAS.)
Obtained Baseline Mammogram | 137 | 133 | 151
Completed | 168 | 162 | 187
Not Completed | 0 | 0 | 0
Period: Year 1: Post Randomization Mammograms
Arm/Group | CEE Pill, Active Progesterone | Estradiol Patch, Active Progesterone | Placebo
Started | 168 (Consented to MDBHAS) | 162 (Consented to MDBHAS) | 187 (Consented to MDBHAS)
Obtained Mammogam | 136 (Obtained post-randomization mammogram) | 123 (Obtained post randomization mammogram) | 148 (Obtained post randomization mammogram)
Completed | 168 | 162 | 187
Not Completed | 0 | 0 | 0
Period: Final: Year 3 or 4 Post-randomization
Arm/Group | CEE Pill, Active Progesterone | Estradiol Patch, Active Progesterone | Placebo
Started | 168 (Consented to MDBHAS) | 162 (Consented to MDBHAS) | 187 (Consented to MDBHAS)
Obtained Year 3 or 4 Mammogram | 143 | 139 | 151
Completed | 168 | 162 | 187
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Population with mammographic density data from at least one time point during study.
Groups:
- Total: Total of all reporting groups
Arm/Group | CEE Pill, Active Progesterone | Estradiol Patch, Active Progesterone | Placebo | Total
Number analyzed (Participants) | 155 | 154 | 179 | 488
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (2.7) | 52.8 (2.5) | 52.6 (2.4) | 52.7 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 154 | 179 | 488
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: BIRADS Breast Density
Description: Breast density prior to randomization. Frequency of the BIRADS category according to randomization status. BIRADS is a 1-4 category of breast density as assessed by a radiologist. 1= most fatty and least dense, while 4=most dense.
Time Frame: Baseline (Prior to Randomization)
Population: Women with mammograms are included.
Measure: Number; unit: participants
Arm/Group | CEE Pill, Active Progesterone | Estradiol Patch, Active Progesterone | Placebo
Number analyzed (Participants) | 137 | 133 | 151
participants
  BIRADS 1 | 9 | 9 | 15
  BIRADS 2 | 42 | 48 | 53
  BIRADS 3 | 79 | 65 | 77
  BIRADS 4 | 7 | 11 | 6

2. Primary Outcome: BIRADS Breast Density
Description: Frequency of the BIRADS category 1 year after randomization. BIRADS is a 1-4 category of breast density as assessed by a radiologist. 1= most fatty and least dense, while 4=most dense.
Time Frame: Year 1
Population: Women with mammograms 1 year after randomization
Measure: Number; unit: participants
Arm/Group | CEE Pill, Active Progesterone | Estradiol Patch, Active Progesterone | Placebo
Number analyzed (Participants) | 136 | 123 | 148
participants
  BIRADS 1 | 10 | 9 | 17
  BIRADS 2 | 47 | 44 | 54
  BIRADS 3 | 74 | 67 | 70
  BIRADS 4 | 5 | 3 | 6

3. Primary Outcome: BIRADS Breast Density
Description: Frequency of the BIRADS category 3-4 years after randomization. BIRADS is a 1-4 category of breast density as assessed by a radiologist. 1= most fatty and least dense, while 4=most dense.
Time Frame: Latest (Year 3 of 4)
Population: Women with mammograms 3-4 years after randomization
Measure: Number; unit: participants
Arm/Group | CEE Pill, Active Progesterone | Estradiol Patch, Active Progesterone | Placebo
Number analyzed (Participants) | 143 | 139 | 151
participants
  BIRADS 1 | 9 | 10 | 18
  BIRADS 2 | 61 | 54 | 70
  BIRADS 3 | 68 | 66 | 55
  BIRADS 4 | 5 | 9 | 8

4. Secondary Outcome: Abnormal Mammogram/Biopsy
Description: Abnormal mammogram requiring additional imaging modality such as MRI or ultrasound, or a breast biopsy. Information obtained from mammography reports.
Time Frame: baseline to 3 years
Population: Women with mammography reports
Measure: Count of Participants; unit: Participants
Arm/Group | CEE Pill, Active Progesterone | Estradiol Patch, Active Progesterone | Placebo
Number analyzed (Participants) | 155 | 151 | 174
Participants | 50 | 63 | 55

ADVERSE EVENTS:
Time Frame: baseline through 4 years.
Description: There were no adverse events related to the ancillary mammographic density study.
Arm/Group | CEE Pill, Active Progesterone | Estradiol Patch, Active Progesterone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/168 | 0/162 | 0/187
Other Adverse Events (participants affected / at risk) | 0/168 | 0/162 | 0/187

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No